CLINICAL TRIAL: NCT06528834
Title: Coronary Angiographic Assessment of Hearts Donated for Transplantation Declined on the Grounds of Visible/Palpable Coronary Artery Disease at the Time of Retrieval
Brief Title: Coronary Artery Disease in Hearts Donated for Transplantation
Status: Not yet recruiting | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 332977
Record Dates: First submitted 2024-07-26; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure
Keywords: heart transplantation; coronary artery disease; coronary angiography
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In spite of recent initiatives, in particular, the introduction into clinical practice of donation after circulatory death (DCD), there is a persistent mismatch between the demand for donor hearts for transplantation and their supply [1]. This mismatch is accentuated by the relatively low rate of utilisation of hearts donated for transplantation, i.e. the proportion of organs transplanted divided by the number of donations. In the UK between 2016 and 2018 this ranged from 25.7 to 30.8% [2]. For the year 2022/23, a total of 207 heart transplants (DBD and DCD) were performed out of 1429 donations giving a utilisation rate of 14.5% [3].

The rigorous assessment of donor heart quality prior to, and during donor organ retrieval, which is a crucial determinant of recipient outcome, accounts for the low utilisation rate. In both the donation after brain(stem) death (DBD) and DCD settings, pre-retrieval echocardiography is the principal method of anatomical and functional assessment. In the DCD setting, where normothermic organ perfusion (either in situ or ex situ) is mandatory to restore myocardial function, additional functional and biochemical assessments are available.

In addition to recipient risk factors, donor age and comorbidity burden continue to limit the applicability and effectiveness of heart transplantation. Older donors are both associated with an increased comorbidity burden and prevalence of coronary artery disease (CAD). Donor-transmitted CAD is of particular concern due to the significant association with early graft dysfunction when multi-vessel disease is present [4,5]. Guidelines recommend that donor hearts with obstructive CAD in any major coronary artery be declined for transplantation [4]. However, there is evidence that single vessel CAD neither alters short- nor long term recipient prognosis [6]. The short and long term risks to the recipient of donor heart CAD needs to be carefully evaluated in relation to the risk of a transplant candidate remaining on the waiting list [7,8].

None of the methods currently available in the UK for the assessment of potential heart donors allows adequate characterisation of coronary artery disease (CAD). Instead, retrieval surgeons place a heavy reliance on an indirect assessment of CAD, i.e. direct visualisation and palpation of the large epicardial coronary arteries with the aim of identifying occlusive lesions. The discovery of such lesions is the justification for declining a donor organ otherwise deemed to be suitable for transplantation.

In other countries, access to coronary artery imaging prior to heart donation is an established option, where indicated. Indeed, the Association of Organ Procurement Organizations Consensus Statement, supported by the Society of Critical Care Medicine and the American College of Chest Physicians recommends coronary angiography in all older donors (>40 years) and in younger patients with risk factors for CAD.

In the proposed study we seek to perform coronary angiography at Harefield Hospital on donated hearts where our retrieval team has declined the organ solely on the grounds of visible/palpable CAD. In so doing we aim to better understand the diagnostic utility of the assessment method. An internal audit of heart retrieval has revealed that of the donated hearts offered to Harefield since 2020 between 8 to 13 are declined per annum on the grounds of visible/palpable coronary artery disease, i.e. approx. 10 per annum. Assuming a study enrolment rate of 1:3 of donated hearts with CAD identified at the time of retrieval, we therefore anticipate that this study will take 36 months to complete. This investigation forms part of a broader research/service improvement initiative which aims to not only enhance the assessment of CAD in potential donors but also to better understand the pathogenesis of CAD in heart transplant recipients. The ultimate goals are to reduce the risks associated with transplantation and increasing donor organ availability. We propose to initiate this investigation as a single centre study but would welcome the participation of other UK centres who would like to collaborate.

We believe this research initiative is well aligned with the strategic objectives of the NHS BT Business Plan 2022-23 [9].

1. Hsich E. Circ. Heart. Fail. 2016 Apr. 9(4) e002679.
2. Rushton and Hogg March 2019 NHSBT/CAG, CHARH(19)25.
3. NHS-BT Annual Activity Report:Section 7, Cardiothoracic activity. 2022-23.
4. Ivanes F et al. Int J Cardiol. 2019 277;71-8.
5. Kotloff RM et al. Crit Care med. 2015;43:1291-325.
6. Dorent et al. Arch. Cardiovasc. Dis. 2018;111:126-39.
7. Kilic A et al. J Thorac Dis. 2014;6:1097-104.
8. Estevz-Loureiro R et al. Transplant. Proc. 2010;42:2987-91.
9. NHS BT Business Plan 2022-23, July 2022.

DETAILED DESCRIPTION:
STUDY RATIONALE AND RISK/BENEFIT ANALYSIS This investigation forms part of a broader research/service improvement initiative which aims to not only improve the assessment of CAD in potential donors but also to better understand the pathogenesis of CAD in heart transplant recipients. The ultimate goals are to reduce the risks associated with transplantation and increase donor organ availability. We propose to initiate this investigation as a single centre study but would welcome the participation of other UK centres who would like to collaborate.

We believe this research initiative is well aligned with the strategic objectives of the NHS BT Business Plan 2022-23, in particular, i) reducing harm to patients (recipients) and ii) achieving the 4-5 year target of higher deceased donor transplant activity by 41.9% [9].

MANAGEMENT OF POTENTIAL STUDY RISKS We have not identified any incremental risks associated with the retrieval and transport of the donated heart beyond those associated with a conventional donor heart retrieval procedure. We are satisfied that suitable arrangements have been made for the appropriate labelling and secure storage of the heart donated for research prior to angiography. We believe the risk of disclosure of donor or recipient identify will be minimised by pseudoanonymisation and the application standard Trust research procedures. Angiography will be performed by an experienced interventional cardiologist. Radiation exposure to clinical personnel during the angiography procedure will be controlled using standard measures.

STUDY OBJECTIVES PRIMARY OBJECTIVE Determination of whether there is discordance between visualisation/palpation and coronary artery angiography for the diagnosis of coronary artery disease.

SECONDARY OBJECTIVES N/a

Prerequisites for commencement of the study include approvals from:

The Research, Innovation and Novel Technologies Advisory Committee (NHSBT) A Research Ethics Committee. Both of these requirements have been fulfilled.

Prerequisites for study enrolment are that:

* the donation centre should be 'within scope' (i.e. holding a suitable HTA licence compatible with organ retrieval for research purposes within the INOAR scheme).
* the donor's family have provided generic consent for the use of untransplantable organs for research purposes.
* the heart is deemed untransplantable on the grounds of the visualisation/palpation of coronary heart disease at the time of retrieval.
* the untransplantable heart is not deemed suitable for valve homograft/patch retrieval
* the untransplanable heart is not allocated to alternative research studies through the INOAR scheme.

If all these criteria are fulfilled and confirmed enrolment may commence. The cardiothoracic retrieval team will give priority to the retrieval of any organs destined for transplantation. The donated heart will be retrieved using the conventional Donation after Brain(stem) Death (DBD) method irrespective of whether the heart was initially offered through the DBD or Donor Circulatory Death (DCD) pathways. The packaging will be labelled using a pseudoanonymised code. The donated heart will be transported to Harefield Hospital by the retrieval team and will be placed within a designated organ storage fridge within the operating theatre facility. Within 24 hours, the interventional cardiologist will perform contrast coronary angiography. After the study procedure, the heart will be made available for further research studies (if appropriate). Alternatively, it will be submitted to disposal using an approved method.

TREATMENT AND RATIONALE Treatment does not feature in the study design. The only proposed intervention is coronary angiography of hearts deemed untransplantable at the time of retrieval on the grounds of visible/palpable coronary artery disease.

ELIGIBILITY CRITERIA INCLUSION CRITERIA Adult hearts donated for transplantation in UK centres attended by the Harefield Retrieval Team yet deemed untransplantable because of visible/palpable coronary artery disease.

Donation centre holds HTA research licence (making the donation of organs for research possible under the INOAR scheme).

EXCLUSION CRITERIA Donation centre does not hold appropriate research licence Donor's family decline to offer generic consent to the use of donated organs for research purposes.

Logistic issues preventing study enrolment.

DISCONTINUATION/WITHDRAWAL OF PARTICIPANTS AND STOPPING RULES N/a. SUBJECT/PATIENT RECRUITMENT PROCESS This will occur through establish transplantation procedures as detailed in 6.1.

STUDY PROCEDURES Left and right coronary artery angiography using standard catheters, radio-opaque dye, in a catheter laboratory at Harefield Hospital.

(We recognise there will be no dye wash-out as occurs during a conventional procedure in a beating heart. If necessary, crystalloid solution will be used to achieve a similar effect).

INFORMED CONSENT Generic consent for the use of untransplantable organs for research purposes is currently sought from the donor's family by the Specialist Nurse in Organ Donation (see attached form).

RANDOMISATION PROCEDURE N/a, single arm study.

EMERGENCY UN-BLINDING N/a STUDY ASSESSMENTS SCREENING ASSESSMENTS No screening assessments are planned.

BASELINE ASSESSMENTS The only relevant baseline assessment is direct visualisation/palpation of the coronary arteries at the time of retrieval of the donated heart.

TREATMENT PROCEDURE Not applicable.

SUBSEQUENT ASSESSMENTS Within 24 hours of retrieval, the donated heart will undergo left and right coronary artery angiography. This procedure will be performed in the catheter laboratory by an experienced Interventional Cardiologist.

SUMMARY CHART OF STUDY ASSESSMENTS Only one procedure will be performed per enrolment within 24 hours of retrieval of the heart donated for research purposes.

METHODS Laboratory Procedures N/a Radiology or any other procedure(s) The study does not entail ionising radiation exposure to a patient. Radiation exposure to clinical staff will be controlled using standard IRMER recommendations.

Is ARSAC licence required? No. Techniques and Interventions Coronary angiography.

Tools Standard left and right heart coronary artery catheters, radio-opaque dye within a catheter laboratory.

Study Drugs N/a.

DEFINITION OF THE END OF STUDY Completion of angiography procedure on the 10th donated heart enrolled in the study followed by data analysis by the designated statistician.

SAFETY REPORTING DEFINITION N/a RECORDING ADVERSE EVENTS (AES)

N/a REPORTING OF SAES TO THE SPONSOR AND THE REC THE TYPE AND DURATION OF THE FOLLOW-UP OF SUBJECT AFTER AES

N/a

PREGNANCY N/a

ANNUAL PROGRESS REPORTS (APRS) The Chief Investigator will prepare the APR for the study. It will be reviewed by the RO and sent to the REC by the CI within 30 days of the anniversary date on which the favourable opinion was given by the REC, and annually until the study is declared ended. A copy of the report will be provided to regulatory stakeholders.

REPORTING URGENT SAFETY MEASURES N/a

DATA MANAGEMENT AND QUALITY ASSURANCE CONFIDENTIALITY All data will be handled in accordance with the Data Protection Act (2018), NHS Caldecott Principles, The UK Policy Framework for Health and Social Care Research, and the condition of the REC approval.

The Case Report Forms (CRFs) will not bear the subject's name or other personal identifiable data. The subject's study Identification Number (ID), will be used for identification.

DATA COLLECTION TOOL Case Report Forms (CRF) will be designed by the CI and the final version will be reviewed and discussed with the study Sponsor. All data will be entered legibly in black ink with a ball-point pen. If the Investigator makes an error, it will be crossed through with a single line in such a way to ensure that the original entry can still be read. The correct entry will then be clearly inserted. The amendment will be initialled and dated by the person making the correction immediately. Overwriting or use of correction fluid will not be permitted.

It is the Investigator's responsibility to ensure the accuracy of all data entered and recorded in the CRFs. The Delegation of Responsibilities Log will identify all study personnel responsible for data collection, entry, handling and managing the database.

The research data will take the form of a pseudoanonymised angiography report, (bearing the ID reference number) provided by the Interventional Cardiologist, of standardised format, with the inclusion of selected angiographic images/videos where appropriate. This information will be compared with the summary report provided by the retrieval surgeon. The custodianship of the research data will be the responsibility of the research nurse.

DATA HANDLING AND ANALYSIS Software: standard coronary angiographic software will be employed for analysis and static and videographic image generation. Reports will be written using Microsoft Word on a Trust computer.

Data quality will be assured by cross referencing to the date of the retrieval procedure.

Research data will be stored on a secure Trust computer with an automated data back-up facility to ensure data security.

Data analysis will be performed by Rachel Hogg, Senior Statistician, NHS BT.

13.4 ARCHIVING ARRANGEMENTS The study documents (including the Study Master File (SMF), Case Report Forms (CRFs), Informed Consent Forms along with the study database) will be kept for a minimum of five years. They will be stored in locked offices within the Royal Brompton and Harefield Hospitals. The CI is responsible for the secure archiving of study documents. The study database will also be kept electronically on the RB&HFT computer network, for a minimum of five years.

The approved repository for longer retention of local materials for studies that involve RB&H patients is Box-It Storage UK. The study documentation will be prepared for archiving by the research team in line with the Research Office Archiving SOP and the transfer will be arranged by the Research Office.

STATISTICAL DESIGN

SAMPLE SIZE AND RECRUITMENT

Ideally, we would have liked to increase the number of donated hearts enrolled in this study. However, there are logistic challenges associated with recruitment and there is competition for such organs for the purposes of homograft valve retrieval and for other research studies.

An internal audit of heart retrieval has revealed that of the donated hearts offered to Harefield since 2020 between 8 to 13 are declined per annum on the grounds of visible/palpable coronary artery disease, i.e. approx. 10 per annum. Assuming a study enrolment rate of 1/3 of donated hearts with CAD identified at the time of retrieval, we therefore anticipate that this study will take 36 months to complete.

Consequently, the endpoints of the proposed study and sample size are not intended to be powered for statistical inference. Instead, the intention is to support or refute a reasonable assurance of the validity of direct visualisation/palpation for the detection of CAD.

Discordance between the diagnosis of coronary artery disease at the time of retrieval and the angiography data (false positive) would be a cause of concern that would provide 'real-world' evidence of the need for coronary artery imaging in organ donors prior to retrieval, where indicated. Rachel Hogg, Senior Statistician, BHS BT, has kindly provided advice concerning study design and has agreed to assist with the data analysis.

ENDPOINTS Primary endpoints The goal of this study is perform coronary angiography on hearts which were retrieved by our transplant team and were declined for transplantation solely on the grounds of visible/palpable (i.e. manual examination) coronary artery disease. In so doing, we aim to better understand whether the current assessment method is reliable. Thus the primary endpoint is discordance between the two diagnostic methods.

Secondary endpoints N/a

STATISTICAL ANALYSIS PLAN See above

Primary endpoint analysis As the study is not powered for detailed statistical inference, data analysis will be of a descriptive nature.

Secondary endpoint analysis N/a

RANDOMISATION N/a INTERIM ANALYSIS (IF APPLICABLE) N/a OTHER STATISTICAL CONSIDERATIONS N/a 15. COMMITTEES INVOLVED IN THE STUDY NHS Organ Donation and Transplantation, Research, Innovation and Novel Technologies Advisory Group (RINTAG) have reviewed the proposed application and given a favourable opinion.

The Lead Clinician for Organ Donation for the UK, Dr Dale Gardiner, has also been informed of our intention to submit this research proposal and is supportive of it, in principle.

Favourable IRB approval was also obtained as detailed above.

MONITORING AND AUDITING The requirement for study monitoring or audit will be based on the internal Research Office risk assessment procedure and applicable Standard Operating Procedures (SOPs). It is the responsibility of the RO to determine the monitoring risk assessment and explain the rationale to the study research team.

Study monitoring and/or audit will be discussed with the CI before arrangements are made to conduct the visit.

DIRECT ACCESS TO SOURCE DATA The Investigator(s)/institution(s) will permit study-related monitoring, audits, REC review, and regulatory inspection(s), providing direct access to source data/documents.

ETHICS AND REGULATORY REQUIREMENTS The Sponsor will ensure that the study protocol, Patient Information Sheet (PIS), Informed Consent Form (ICF), GP letter and submitted supporting documents have been approved by the Health Research Authority (HRA) which includes Research Ethics Committee (REC) approval if applicable, prior to any patient recruitment taking place. The protocol and all agreed substantial protocol amendments, will be documented and submitted for HRA approval prior to implementation.

Before site(s) can enrol patients into the study confirmation of capacity and capability must be issued by the institution hosting the trial (unless HRA specifically has confirmed in the HRA approval letter that this is not required). It is the responsibility of the PI at each site to ensure that all subsequent amendments gain the necessary approvals by the participating site. This does not affect the individual clinician's responsibility to take immediate action if thought necessary to protect the health and interest of individual patients.

Within 90 days after the end of the study, the CI will ensure that the REC is notified that the study has finished. If the study is terminated prematurely, those reports will be made within 15 days after the end of the study.

The CI will supply a final summary report of the clinical study to the REC and the Sponsor in parallel within one year after the end of the study.

FINANCE

* 8,300 has been allocated from an internal Trust research account for the proposed study. This is sufficient to cover:
* 1,500 RINTAG application fee (which covers the first 12 months of the study).
* 600 (2 x £300 annual renewal fee for the above) to enable the study to run for 36 months.
* 6,000 (10 x £600 per angiography investigation - fully funded angiography - costs kindly provided by the Divisional Interventional Lead, Cardiology).

On this basis, sufficient funds are available for the enrolment of 10 donated hearts with a contingency of £200.

There will be no incremental transport costs as our Transplant Retrieval Team will be attending the donation centre in the course of their normal duties.

INSURANCE AND INDEMNITY N/a PUBLICATION POLICY Data ownership rights will reside with the host institution. STATEMENT OF COMPLIANCE The trial will be conducted in compliance with the protocol, Sponsor's Standard Operating Procedures (SOPs), GCP and the applicable regulatory requirement(s).

The study conduct shall comply with all relevant laws of the UK country in which the study site is located including but not limited to, the Human Rights Act 1998, the Data Protection Act 2018, and with all relevant guidance relating to medicines and clinical studies from time to time in force including, but not limited to, the ICH GCP, the World Medical Association Declaration of Helsinki entitled 'Ethical Principles for Medical Research Involving Human Subjects' (2008 Version), the UK Policy Framework for Health and Social Care Research.

This study will be conducted in compliance with the protocol approved by HRA and according to RGF standards. No deviation from the protocol will be implemented without the prior review and approval of the Sponsor and HRA except where it may be necessary to eliminate an immediate hazard to a research subject. In such case, the deviation will be reported to the Sponsor and the REC as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

Hearts donated for transplantation which are retrieved by the Harefield Hospital retrieval team which are deemed untransplantable on the grounds of visible or palpable coronary artery disease of the epicardial arteries at the time of retrieval.

-

Exclusion Criteria:

Absence of family consent to retrieve untransplantable heart for research purposes

Logistic challenges

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hearts donated for transplantation which are retrieved by the Harefield Hospital retrieval team
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Discordance | 3 years
  The goal of this study is perform coronary angiography on hearts which were retrieved by our transplant team and were declined for transplantation solely on the grounds of visible/palpable (i.e. manual examination) coronary artery disease. In so doing, we aim to better understand whether the current assessment method is reliable. Thus the primary endpoint is discordance between the two diagnostic methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Brompton and Harefield Hospital NHS Trust, London, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only aggregate anonymised data will be shared.